CLINICAL TRIAL: NCT01593215
Title: Randomized Study of Yohimbine Treatment for Type 2 Diabetes Patients Carrying a Specific Genetic Risk Variant
Acronym: YOH1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anders Rosengren, MD PhD (Other)
Collaborators: Region Skane (Other); Lund University (Other)
Responsible Party: Sponsor-Investigator, Anders Rosengren, MD PhD, MD PhD, Region Skane
Organization: Region Skane (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-018604-85
Record Dates: First submitted 2012-05-03; First posted 2012-05-08 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes
Keywords: genetics; type 2 diabetes; insulin secretion
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Yohimbine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo first then yohimbine (Active Comparator): placebo first, then yohimbine
  Interventions: Drug: Yohimbine
- Yohimbine first then placebo (Active Comparator): Yohimbine first then placebo
  Interventions: Drug: Yohimbine

INTERVENTIONS:
Drug: Yohimbine — Yohimbine capsule

SUMMARY:
The investigators have recently discovered a genetic variant in an adrenergic receptor that leads to increased risk for type 2 diabetes. The investigators have also seen that blockers of that receptor improves impaired insulin secretion in animals. The investigators will now test the blocker in patients with type 2 diabetes with or without the risk variant in an effort to make diabetes treatment more individualized.

DETAILED DESCRIPTION:
We have recently discovered a genetic variant in an adrenergic receptor that leads to increased risk for type 2 diabetes. We have also seen that blockers of that receptor improves impaired insulin secretion in animals. We will now test the blocker in patients with type 2 diabetes with or without the risk variant in an effort to make diabetes treatment more individualized. Patients will receive two different doses of the blocker and the effect will be measured with oral glucose tolerance tests. The study is a randomized placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* informed consent
* age 18-70, for females only postmenopausal

Exclusion Criteria:

* heart disease
* anxiety disorder
* antidiabetic treatment other than metformin
* adrenergic blockers
* ulcus
* allergy to any component in the capsules

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Rosengren, MD PhD, Principal Investigator — Region Skane
Locations (1):
- Skanes Universitetssjukhus, Malmo, Skåne County, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First Then Yohimbine: Placebo first, then 2 weeks washout and then yohimbine
- Yohimbine First Then Placebo: Yohimbine first, 2 weeks washout and then placebo
Period: Overall Study
Arm/Group | Placebo First Then Yohimbine | Yohimbine First Then Placebo
Started | 25 | 25
Completed | 24 | 25
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo First Then Yohimbine: placebo first
  Yohimbine: Yohimbine capsule
- Yohimbine First Then Yohimbine: Yohimbine first and then placebo
- Total: Total of all reporting groups
Arm/Group | Placebo First Then Yohimbine | Yohimbine First Then Yohimbine | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (8) | 60 (7) | 60 (8)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 20 | 22 | 42
Region of Enrollment [Number; unit: participants]
  Sweden | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Insulin Secretion
Description: insulin secretion will be measured (nMole) in response to an oral glucose tolerance test. Patients will receive the capsules 1 h before the glucose test, and the insulin levels 30 minutes after the oral glucose will be used as a primary outcome measure. The insulin levels at the highest tolerated dose of yohimbine will be used.
Time Frame: 30 minutes after oral glucose
Measure: Mean (95% Confidence Interval); unit: % increase of Ins30
Groups:
- Placebo: placebo
  Yohimbine: Yohimbine capsule
- Yohimbine: Yohimbine
  Yohimbine: Yohimbine capsule
Arm/Group | Placebo | Yohimbine
Number analyzed (Participants) | 49 | 49
% increase of Ins30 | 5 [-13 to 20] | 29 [5 to 52]

2. Secondary Outcome: Glucose
Description: Plasma glucose will be measure (mMole) in response to an oral glucose tolerance test. Patients will receive the capsules 1 h before the glucose test, and the glucose levels 30 minutes after the oral glucose will be used as a secondary outcome measure. The glucose levels at the highest tolerated dose of yohimbine will be used.
Time Frame: 30 minutes after oral glucose
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo | Yohimbine
Serious Adverse Events (participants affected / at risk) | 0/49 | 1/49
Other Adverse Events (participants affected / at risk) | 0/49 | 6/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | Yohimbine (N=49)
Transitory ischemic attack (Vascular disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | Yohimbine (N=49)
Anxiety (Psychiatric disorders) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No